CLINICAL TRIAL: NCT04742426
Title: Does the Choice of Personal Protective Equipment Affect Team Performance During Medical Emergencies? Simulation-Based Randomised Controlled Trial
Brief Title: Personal Protective Equipment Affect Team Performance During Medical Emergencies
Acronym: PPE-TEAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Roman Sýkora (Other)
Responsible Party: Sponsor-Investigator, Roman Sýkora, assistant professor, Charles University, Czech Republic
Organization: Charles University, Czech Republic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PPE-TEAM
Record Dates: First submitted 2021-01-20; First posted 2021-02-08 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Safety Issues; Communication; Cardiopulmonary Arrest
Keywords: Personal Protective Equipment; Simulation Study; Cardiopulmonary Resuscitation; Non-Technical Skills
MeSH Terms: conditions — Communication; Heart Arrest

STUDY DESIGN:
Intervention Model Description: single-center, randomized (1:1), parallel-group, simulation study
Who Masked: Outcomes Assessor
Masking Description: Blinding of participants and researchers involved in the experiment is not possible. Only the outcome assessor and data analyst is kept blinded to the allocation of subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WHO group (Active Comparator): minimal setting of personal protective equipment (COVID 19) recommended by WHO
  Interventions: Other: WHO recommended PPE
- Super-safe setup (Experimental): maximal super-safe setup of personal protective equipment
  Interventions: Other: Super-safe setup

INTERVENTIONS:
Other: WHO recommended PPE — Uses polycarbonate safety spectacles, fluid-resistant (Type IIR) surgical mask and disposable surgical gown. No head or foot cover.
  Arms: WHO group
Other: Super-safe setup — Uses surgical cap, FFP3 respirator covered by surgical mask, face shield, whole-body suit (Tyvec), 3 pairs of gloves typed to suit sleeves and disposable foot cover.
  Arms: Super-safe setup

SUMMARY:
Safety of healthcare professionals working in high-risk environments is of upmost importance. Personal protective equipment (PPE) may affect the performance of individuals and teams by altering their senses, manual skills and ability to communicate. Current guidelines offer flexibility in terms of which specific PPE components can safely be used. Yet, in some organisations, healthcare workers become used to using PPE well above the recommended standards (termed further in text as super-safe setup, SSS). Impact of this PPE policy on team performance and in turn to patient safety is unknown. The investigators hypothesise that SSS, as compared to WHO PPE standard, would negatively impact team performance and patient outcomes in a simulated crisis scenario.

DETAILED DESCRIPTION:
Safety of healthcare professionals working in high-risk environments is of upmost importance. Personal protective equipment (PPE) may affect the performance of individuals and teams by altering their senses, manual skills and ability to communicate. Current guidelines (WHO, UK, ECDC) offer flexibility in terms of which specific PPE components can safely be used. Yet, in some organisations, healthcare workers become used to using PPE well above the recommended standards (termed further in text as super-safe setup, SSS). Impact of this PPE policy on team performance and in turn to patient safety is unknown. The investigators hypothesise that SSS, as compared to WHO PPE standard, would negatively impact team performance and patient outcomes in a simulated crisis scenario.

Methods Design: prospective, open, randomised, controlled, parallel group trial, fully compliant with CONSORT guidelines with extension for simulation studies.

Study subjects: doctors and nurses routinely working in intensive care, written prospective informed consent Setting: High-fidelity simulation centre, Third Faculty of Medicine, Charles University in Prague

PPE tested

* WHO group (CONTROL): uses polycarbonate safety spectacles, fluid-resistant (Type IIR) surgical mask and disposable surgical gown. One pair of gloves. No head or foot cover.
* SSS group: Uses surgical cap, FFP3 respirator covered by surgical mask, face shield, whole-body suit (Tyvec), 3 pairs of gloves typed to suit sleeves and disposable foot cover

Study procedures: Teams consisting of one doctor and two nurses will be recruited. The purpose of the study will be explained to them as a part of consent procedure, but details of evaluation and scenarios will remain undisclosed. All team members will obtain standardized educational materials focused on the solution of airway management and non-shockable rhythm of sudden circulatory arrest in a critically ill patient.

* Introduction to simulation centre and baseline team performance measurement: On the study day the teams will undergo a standardised introduction to simulation centre and perform a mock scenario without PPE apart from gloves and simple surgical masks. The same parameters will be measured for mock scenario as for the test scenario.
* Test scenario: This will be a COVID-19 patient on mechanical ventilator who suddenly loses airways and develops profound hypoxia progressing to cardiac arrest. Team will be wearing PPE according to their study group allocation at the beginning of the scenario.

Outcomes:

• Primary outcome: Non-technical team performance measured as TEAM score and adjusted to baseline team performance

• Secondary outcomes: Quality of CPR and work according to guidelines

• Exploratory qualitative objective: physiological functions of team members and self-reported confidence defined on visual analogue scale

Outcome assessment methods: Performance indices will be observed by two independent, trained assessors. Both assessors will have access to video recordings of scenarios and software recordings. The final score will be an arithmetic mean of the scores of two observers. Inter-rater variability will be calculated and reported.

Sample size calculation and statistics: According to [ref] the TEAM performance score was 3.3±0.7 (mean±standard deviation). Therefore, n=22 (i.e. 11 teams per group) gives 80% probability of detecting at p<0.05 (two sided) 25% difference of TEAM scores between groups. Primary outcome will be calculated by two sided Student t-test. Time-to-event outcomes will be compared using Kaplan-Meier curves and Wilcoxon test.

Dissemination plan and implementation: Data will be published in a peer-reviewed journal. The results have the potential to influence hospital hygiene policies as well as choices made by individual healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Medicine (EM) and Anesthesiology and Critical Care (ACC) physicians
* Emergency Medicine (EM) and Anesthesiology and Critical Care (ACC) nurses
* Preparation and study of sent educational materials
* Fulfillment of the whole complete simulation

Exclusion Criteria:

* Not giving or withdrawal of the informed consent
* Not willing to participate
* Incomplete data acqusition

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
The Team Emergency Assessment Measure score (TEAM score) | During the intervention
  The TEAM questionaire will be used and will address following items: 1) the team leader let the team know what was expected of them through direction and command, 2) the team leader maintained a global perspective, 3) the team communicated effectively, 4) the team worked together to complete tasks in a timely manner, 5) the team acted with composure and control, 6) the team morale was positive, 7)the team adapted to changing situations, 8) the team monitored and reassessed the situation, 9) the team anticipated potential actions, 10) the team prioritized tasks, 11) the team followed approved standards/guidelines and 12) the global score. The TEAM items 1 - 11 will be rated using a five-point scale (range 0-4; 0 never/hardly ever, 1 seldom, 2 about as often as not, 3 often, 4 always/nearly always). The item 12 (global score) - the overall performance will be rated on scale from 1 to 10 (best). The mean for each item will be calculated.

SECONDARY OUTCOMES:
Time to first chest compression | During the intervention
  Time to first chest compression from the start of the scenario will be measured in seconds. Time will be obtained from the software recording of the simulator as time to first compression to reach depth at least 5cm.
Time to first epinephrine dose administration | During the intervention
  The time to to first epinephrine dose administration (seconds) will be measured by observer and checked from the simulator recording.
Time to first effective breath after reintubation | During the intervention
  The time to perform the first effective breath (tidal volume of at least 400ml) after reintubation will be measured in seconds . The time will be obtained from the software recording of the simulator.
Chest compression frequency | During the intervention
  Average chest compression rate (per minute) will be calculated from from the software recording of the simulator. In addition, the percentage of time out of the total compression time, when the frequency of 100-120 per minute was reached, will be measured.
Chest compression depth | During the intervention
  Average chest compression depth (cm) will be obtained from the software recording of the simulator. In addition, the percentage of compressions reaching a depth of 5 - 6 cm from the total number of compressions will be calculated.

OTHER OUTCOMES:
Blood pressure of team members | During the intervention
  Blood pressure of all the team members will be monitored in two minutes intervals throughout the simulation.
Heart rate of team members | During the intervention
  Heart rate of all the team members will be monitored continuously throughout the simulation.
Breathing frequency | During the intervention
  The breathing frequency will be measured in all the team members in resting condition and than continuously throughout the simulation.
Body temperature of team members | Immediately after the intervention
  Blood temperature of all the team members will be measured in resting condition and at the end of the simulated scenario.
Self assessment of the team performance | Immediately after the intervention
  The self assessment of the team performance by all the teams members will be obtained. The score will be evaluated by the team members from one to ten points, where ten points indicate the best possible performance.

CONTACTS AND LOCATIONS:
Overall Officials: Frantisek Duska, PhD, Study Director — Third Medical Faculty and FNKV University Hospital, Charles University in Prague, Czech Republic

IPD SHARING:
Plan to Share IPD: No
All data, forms, consents and protocols will be provided on reasonable request by investigators.

REFERENCES:
- [Result] Mormando G, Paganini M, Alexopoulos C, Savino S, Bortoli N, Pomiato D, Graziano A, Navalesi P, Fabris F. Life-Saving Procedures Performed While Wearing CBRNe Personal Protective Equipment: A Mannequin Randomized Trial. Simul Healthc. 2021 Dec 1;16(6):e200-e205. doi: 10.1097/SIH.0000000000000540. PMID 33428358
- [Result] Cooper S, Cant R, Porter J, Sellick K, Somers G, Kinsman L, Nestel D. Rating medical emergency teamwork performance: development of the Team Emergency Assessment Measure (TEAM). Resuscitation. 2010 Apr;81(4):446-52. doi: 10.1016/j.resuscitation.2009.11.027. Epub 2010 Feb 1. PMID 20117874